CLINICAL TRIAL: NCT04396795
Title: A Randomized Control, Double-Blind, Placebo Controlled, Multicenter Clinical Trial on Safety and Efficacy of Autologous Platelet-Rich Plasma Injection Treatment for Erectile Dysfunction.
Brief Title: Safety and Efficacy of Autologous Platelet-Rich Plasma for Erectile Dysfunction.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Director of Male Fertility and Andrology, University of Miami, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200373
Record Dates: First submitted 2020-04-03; First posted 2020-05-21 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Erectile Dysfunction
Keywords: ED
MeSH Terms: conditions — Erectile Dysfunction | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP group (Experimental): Participants in this group will receive 2 sessions of autologous PRP penile injection, each administered 1 month apart ± 7 days
  Interventions: Drug: Autologous Platelet Rich Plasma
- Placebo group (Placebo Comparator): Participants in this group will receive 2 sessions of placebo injection, each administered 1 month apart ± 7 days.
  Interventions: Other: Saline solution

INTERVENTIONS:
Drug: Autologous Platelet Rich Plasma — Each injection session will consist of a total of 5 mL PRP infused slowly over a 2-minute period; 2.5 mL each injected to the right and left corpus cavernosum.
  Other Names: PRP
  Arms: PRP group
Other: Saline solution — Each injection session will consist of a total of 5 mL saline solution infused slowly over a 2-minute period; 2.5 mL each injected to the right and left corpus cavernosum
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate changes in vascular parameters and International Index of Erectile Function (IIEF) scores with the administration of Platelet Rich Plasma (PRP) to participants with Erectile Dysfunction (ED)

ELIGIBILITY:
Inclusion Criteria:

1. Be Male
2. Be 30 to 75 years of age (inclusive).
3. Be able to provide written informed consent.
4. Have a diagnosis of ED due to organic origin for at least 6 months prior to consent.
5. Sexually active in a stable, heterosexual relationship of more than three months duration.
6. IIEF-EF score 11-25 at screening (even if taking a single PDE5).
7. Agree to attempt sexual intercourse at least 4 times per month for the duration of the study without being under the influence of alcohol or recreational drugs.
8. Agree to comply with all study related tests/procedures.

Exclusion Criteria:

1. Previous penile surgery of any kind (except circumcision and condyloma removal), such as penile lengthening, penile cancer surgery, penile plication, grafting.
2. Previous history of priapism or penile fracture
3. Abnormal morning serum testosterone level defined as a value lower than 300 ng/dL (±5%) (indicative of untreated hypogonadism), or greater than 1197 ng/dL (±5%).
4. Current or previous hormone usage, other than prescribed testosterone, clomiphene or thyroid medication. (Subjects with prior or current use of hormonal treatment for prostate cancer are also excluded.
5. Psychogenic ED as determined by study investigator.
6. Anatomical (Peyronie's Disease or penile curvature that negatively influences sexual activity) or neurological abnormalities in the treatment area.
7. Patients using Intra Cavernous Injection (ICI)for management of ED
8. Patients with generalized polyneuropathy, or neurological conditions irrespective of cause, such as severe diabetes, multiple sclerosis or Parkinson's disease.
9. Have a serious comorbid illness/condition/behavior that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.
10. History of consistent treatment failure with PDE5 inhibitors for therapy of ED.
11. Any history of significant psychiatric disease, such as bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity. Patients who are currently using Selective Serotonin Reuptake Inhibitor or psychotropic medications.
12. Hemoglobin a1c >9%.

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andia I, Maffulli N. Platelet-rich plasma for managing pain and inflammation in osteoarthritis. Nat Rev Rheumatol. 2013 Dec;9(12):721-30. doi: 10.1038/nrrheum.2013.141. Epub 2013 Oct 1. PMID 24080861
- [Background] Sampson S, Gerhardt M, Mandelbaum B. Platelet rich plasma injection grafts for musculoskeletal injuries: a review. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):165-74. doi: 10.1007/s12178-008-9032-5. PMID 19468902
- [Background] Xie X, Zhang C, Tuan RS. Biology of platelet-rich plasma and its clinical application in cartilage repair. Arthritis Res Ther. 2014 Feb 25;16(1):204. doi: 10.1186/ar4493. PMID 25164150
- [Background] Randelli P, Randelli F, Ragone V, Menon A, D'Ambrosi R, Cucchi D, Cabitza P, Banfi G. Regenerative medicine in rotator cuff injuries. Biomed Res Int. 2014;2014:129515. doi: 10.1155/2014/129515. Epub 2014 Aug 13. PMID 25184132
- [Background] Galliera E, Corsi MM, Banfi G. Platelet rich plasma therapy: inflammatory molecules involved in tissue healing. J Biol Regul Homeost Agents. 2012 Apr-Jun;26(2 Suppl 1):35S-42S. PMID 23648197
- [Background] Nurden AT, Nurden P, Sanchez M, Andia I, Anitua E. Platelets and wound healing. Front Biosci. 2008 May 1;13:3532-48. doi: 10.2741/2947. PMID 18508453
- [Background] Lin G, Shindel AW, Fandel TM, Bella AJ, Lin CS, Lue TF. Neurotrophic effects of brain-derived neurotrophic factor and vascular endothelial growth factor in major pelvic ganglia of young and aged rats. BJU Int. 2010 Jan;105(1):114-20. doi: 10.1111/j.1464-410X.2009.08647.x. Epub 2009 Jun 2. PMID 19493269
- [Background] Apel PJ, Ma J, Callahan M, Northam CN, Alton TB, Sonntag WE, Li Z. Effect of locally delivered IGF-1 on nerve regeneration during aging: an experimental study in rats. Muscle Nerve. 2010 Mar;41(3):335-41. doi: 10.1002/mus.21485. PMID 19802878
- [Background] Werner S, Grose R. Regulation of wound healing by growth factors and cytokines. Physiol Rev. 2003 Jul;83(3):835-70. doi: 10.1152/physrev.2003.83.3.835. PMID 12843410
- [Background] Kushida S, Kakudo N, Morimoto N, Hara T, Ogawa T, Mitsui T, Kusumoto K. Platelet and growth factor concentrations in activated platelet-rich plasma: a comparison of seven commercial separation systems. J Artif Organs. 2014 Jun;17(2):186-92. doi: 10.1007/s10047-014-0761-5. Epub 2014 Apr 20. PMID 24748436

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | PRP Group | Placebo Group
Started | 28 | 33
Completed | 28 | 33
Not Completed | 0 | 0
Period: Month 1
Arm/Group | PRP Group | Placebo Group
Started | 28 | 33
Completed | 26 | 30
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3
Period: Month 3
Arm/Group | PRP Group | Placebo Group
Started | 26 | 30
Completed | 25 | 27
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3
Period: Month 6
Arm/Group | PRP Group | Placebo Group
Started | 25 | 27
Completed | 22 | 24
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRP Group | Placebo Group | Total
Number analyzed (Participants) | 28 | 33 | 61
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [38.5 to 55] | 46 [42 to 56] | 47 [41 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 28 | 33 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 21 | 36
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 23 | 26 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving MCID in IIEF-EF.
Description: Minimal clinically important difference (MCID) is measured by the number of participants who have achieved an increase in International Index of Erectile Function - Erectile Function Subdomain Score (IIEF-EF) based on their Erectile Dysfunction (ED) severity at baseline (an increase of 2 points from baseline for participants with mild ED and an increase of 5 points for participants with moderate ED). MCID in IIEF-EF scores are used to determine treatment efficacy of PRP compared to placebo. IIEF-EF is a 5-item subdomain self- evaluation questionnaire of erectile function with a total score ranging from 0-25 with the higher score indicating better erectile function. This outcome is reported as the number of participants who achieve MCID in each treatment group.
Time Frame: 1 month, 3 month, 6 month
Population: Not all subjects completed all visits due to lost to follow up or did not complete the IIEF questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Group | Placebo Group
Number analyzed (Participants) | 24 | 28
Participants
  Month 1 | 14 | 15
  Month 3: number analyzed (Participants) | 24 | 25
  Month 3 | 10 | 13
  Month 6: number analyzed (Participants) | 20 | 24
  Month 6 | 12 | 10

2. Secondary Outcome: Change in IIEF-EF Scores
Description: IIEF-EF is a 5-item subdomain self-evaluation questionnaire of erectile function. Each item is scored from 0-5 with the total score ranging from 0-25 with the higher score indicating better erectile function.
Time Frame: Baseline up to Month 1, Month 3, and Month 6
Population: Not all subjects completed all visits due to lost to follow up or did not complete the IIEF questionnaire.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PRP Group | Placebo Group
Number analyzed (Participants) | 24 | 28
score on a scale
  Baseline to Month 1 | 4.5 [0 to 8.5] | 2 [-0.5 to 8]
  Baseline to Month 3: number analyzed (Participants) | 24 | 25
  Baseline to Month 3 | 1 [-3 to 7.5] | 2 [-1 to 6]
  Baseline to Month 6: number analyzed (Participants) | 20 | 24
  Baseline to Month 6 | 3.5 [0 to 9.5] | 2 [-2.5 to 7]

3. Secondary Outcome: Change in Doppler Ultrasound Parameters - Peak Systolic Velocity (PSV)
Description: Change in Peak Systolic Velocity (PSV) assessed in cm/sec via ultrasound.
Time Frame: Baseline to Month 6
Population: Not all subjects completed all visits due to lost to follow up.
Measure: Median (Inter-Quartile Range); unit: cm/sec
Arm/Group | PRP Group | Placebo Group
Number analyzed (Participants) | 22 | 24
cm/sec | 0.4 [-9.6 to 15.3] | 1.5 [-3.4 to 14.8]

4. Secondary Outcome: Number of Adverse Events
Description: Incidence of adverse events were reported as all urological and/or reproductive system AEs and all AEs with severity grade 3 or higher. Adverse Events severity was determined using CTCAE v5 criteria.
Time Frame: 24 weeks
Measure: Number; unit: events
Arm/Group | PRP Group | Placebo Group
Number analyzed (Participants) | 28 | 33
events | 1 | 1

5. Secondary Outcome: Number of Participants With an End Diastolic Velocity (EDV) Value Greater Than 0, as Assessed by Penile Doppler Ultrasound at Baseline and Month 6.
Description: Number of participants who had an End Diastolic Velocity (EDV) value of greater than 0, as assessed by penile doppler ultrasound.
Time Frame: Baseline and Month 6
Population: The number of participants analyzed are different in certain rows due to attrition and lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Group | Placebo Group
Number analyzed (Participants) | 28 | 33
Participants
  Baseline | 6 | 11
  Month 6: number analyzed (Participants) | 24 | 26
  Month 6 | 9 | 8

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PRP Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/33
Other Adverse Events (participants affected / at risk) | 1/28 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRP Group (N=28) | Placebo Group (N=33)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 0 (0) — New Penile Plaque

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT04396795/Prot_SAP_000.pdf